CLINICAL TRIAL: NCT02866851
Title: Feasibility Study of Monitoring by Web-application on Cytopenia Related to Chemotherapy
Acronym: BioConnect
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Only one center could be open and the center could not include all patients
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICO-A-2014-12; 2014-A01902-45 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2016-07-21; First posted 2016-08-15 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Monitoring by Web application (Experimental): Patients have to log in a web-application every day (from D5) to indicate their temperature and the presence of gravity sign in case of fever.
  Interventions: Other: Monitoring by Web-application

INTERVENTIONS:
Other: Monitoring by Web-application — Patients have to log in a web-application every day (from D5) to indicate their temperature and the presence of gravity sign in case of fever.
  Other Names: New technology

SUMMARY:
Patients should receive a chemotherapy regimen with an overall risk of febrile neutropenia ≥ 20%. The use of the web-application their will be proposed .

They will be informed of the risk of neutropenia, fever and bleeding which may occur beyond the fifth day of each chemotherapy cycle (to eliminate fevers related to treatment).

The temperature measurement is performed at home by an infrared forehead thermometer provided as part of the study, in a systematic manner once daily at the same time of day and in case of unexplained fatigue or chills.

Before any fever reported to the physician via the web-application (alert), a questionnaire will be completed by the patient to the search for gravity criteria to assess his condition at home. The patient will be hospitalized immediately if it shows signs of severity in order to document the infection and provide intravenous antibiotics adapted to the clinical condition; in the absence of these signs, the patient will make a count to the nearest lab and will receive oral antibiotics if indicated. The subsequent strategy will be defined by the web-application algorithm to optimize the care of patients.

The ability to use a web-application could allow early detection of complications of post-chemotherapy haematological toxicity and offer a taking over guided by a decision-making algorithm managed by the physician.

The aim is to favour the taking over at home.

DETAILED DESCRIPTION:
The hematological toxicity is frequent and sometimes severe complication of chemotherapy used in onco-hematology.

The most frequent is the neutropenia. It is defined by Neutrophils rate lower than 1 Giga/L. The patient can then have a risk of fever or serious infection which requires a hospitalization, an empiric antibiotic therapy and sometimes a dose reduction of chemotherapy which can threaten the patient future. Hospital overall mortality by febrile neutropenia is estimated at 9.5%.

The growth factor allowed to reduce the risk of neutropenia or to shorten the neutropenia. In general, they are suggested in primary prophylaxis for chemotherapy whose risk of febrile neutropenia is superior at 20%.

However, only 20 to 30% of post-chemotherapy fever will be documented. A double and early empiric antibiotic therapy decreases significantly the risk of mortality.

Thrombocytopenia is a less frequent complication than the neutropenia but there is a risk of spontaneous bleeding for the patient when the platelets rate is below 10 Giga/L.

The patient is informed at the beginning of his taking care of the neutropenia risk, fever and hemorrhagic event which can happen at home between two chemotherapies. The patient is in the center of his taking care of and must report quickly all fever or bleeding happening after chemotherapy to evaluate the risk of immediate complication and to propose the appropriate therapeutic strategy. However too many patient with one or two hematological complication during the chemotherapy aren't take care of optimally nor in adapted delay.

The use of a web-application could allow to febrile patient after chemotherapy to benefit of personalized care with a quicker communication of clinical symptoms and blood tests results to the oncologist via this tool.

In practice, patients don't always contact their oncologist in case of fever. On the other hand, the delays for transmission of biological tests at the medical team don't always allow an optimal taking care of and in appropriate delays of hematological toxicity and febrile event of patient during chemotherapy.

The possibility of using a web-application could allow to detect earlier the possible complication of post-chemotherapy hematological toxicity and to suggest a taking care of guided by a decisional algorithm managed by the oncologist. The aim is to privilege the care at home.

The expected benefit for each patient is to have an earlier and adapted care in case of infection and/or bleeding. The use of this web-application could allow, in optimizing the care of chemotherapy-induced neutropenia, to limit the number of hospitalization and the prescription of intravenous antibiotic and to achieve optimally the therapeutic project.

The usual monitoring (oral advice only) would have been proposed at all patient include in this study. It is unlikely that post-chemotherapy fever, neutropenia or thrombocytopenia will supported later than in the usual practice. Therefore it is expected that the use of the web-application will be for the benefit of patient by allowing to detect earlier post-chemotherapy complications and so to propose an optimal take care of for included patients.

Patient must have a chemotherapy schema with a global risk of febrile neutropenia < 20% could use the web-application.

Patients will be informing of the risks of neutropenia, fever and bleeding could happen beyond the 5th day after chemotherapy.

Temperature will be taken at home by an infrared forehead thermometer provided in the study in a systematic once a day at the same time and in case of unusual fatigue or chills.

When a fever is detected by the web-application, a questionnaire will be completed by the patient to find serious symptoms. The aim is to optimize the taking care of patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a histologically proven cancer regardless of the location (solid tumor or not) except brain tumor
2. Patient should receive chemotherapy (any indication) associated with overall risk of neutropenia greater than or equal to 20%
3. Age ≥ 18 years
4. Performance Status ≤ 3
5. Patient with Internet access and an email box
6. Patient affiliated to a social security scheme
7. Patient has given its written consent before any specific procedure for the study

Exclusion Criteria:

1. Symptomatic brain metastases
2. Persons deprived of liberty, under guardianship or under curators
3. dementia, mental impairment or psychiatric illness that may affect the patient's informed consent and / or protocol adherence and monitoring of the test
4. Patient unable to submit the protocol followed for psychological, social, family or geographical reasons
5. Pregnant or breastfeeding
6. Patients at risk of severe neutropenia (Absolute Neutrophils Count <0.1 Giga / L within 7 days prior to inclusion, acute leukemia, auto or allograft)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Patient compliance with the use of the web-application which will be assessed by the number of completed evaluations compared to the theoretical number of filling. | 4 months
The opinion of the patients regarding this application will be assessed through a satisfaction survey completed in the 4th cycle of chemotherapy (3rd cycle for patients receiving 3 CEF100 (Cytoxan-Ellance-Fluorouracil) then Taxotere). | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice DENIS, MD, Principal Investigator — Institut interrégionaL de Cancérologie - LA MANS
Locations (1):
- Institut interregionaL de Cancérologie, Le Mans, France